CLINICAL TRIAL: NCT03016403
Title: A Stepped-Care Intervention to Reduce Disparities in Mental Health Services Among Underserved Lung and Head and Neck Cancer Patients and Their Caregivers
Brief Title: A Stepped Care Intervention to Reduce Disparities in Mental Health Services Among Cancer Patients and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-2621.cc; AD-1511-33395 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2016-12-27; First posted 2017-01-10 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-02

CONDITIONS: Cancer, Lung; Cancer, Head and Neck
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped-Care Intervention (Experimental): Intervention strategies are grounded in evidence-based Cognitive Behavioral Therapy (CBT), that includes stress management and relaxation treatment strategies and coping skills training. Treatment strategies have been adapted from the Transactional Model of Stress and Coping (TMSC), a theoretical model that predicts that individuals who are able to cope and adapt to the stress related to cancer treatment or caregiving will report less psychological distress than those unable to cope.
  Interventions: Behavioral: Stepped-Care Intervention
- Enhanced Usual Care (Active Comparator): Denver Health, St. Mary's and St. Joseph's hospitals provide supportive mental health care for patients such as printed materials, support groups, crisis counseling, and specialized care (e.g., psychiatric medication). Because the amount of usual mental health care that each patient receives varies at each site, the investigators will standardize and monitor the usual care arm across the three sites with an enhanced usual care condition.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Stepped-Care Intervention — The intervention delivered evidence-based CBT and stress management across eight counseling sessions.
  Arms: Stepped-Care Intervention
Behavioral: Enhanced Usual Care — Consists of a list of standard mental health resources offered at the participating hospital, local community, or national non-profit organizations.
  Other Names: Standard of Care
  Arms: Enhanced Usual Care

SUMMARY:
Medically under-served (i.e., low-income, uninsured, underinsured) cancer patients generally encounter significant disparities in accessing care for their mental health needs while undergoing toxic treatments that provide considerable physical and emotional stress. Thus, the investigators propose to adapt evidence-based strategies to a stepped-care intervention model to address the mental health needs of under-served lung cancer (LC) and head and neck cancer (HNC) patients and their caregivers across several levels of symptom severity (e.g., mild, moderate, or severe symptoms of depression and anxiety).

ELIGIBILITY:
1. LC and HNC patients:

   Inclusion Criteria:
   * Newly diagnosed LC and/or HNC (within a month of recruitment date from the date of 1st visit oncology, Ear Nose and Throat (ENT), or radiation clinic visit/consultation upon pathologic tissue diagnosis;
   * LC and/or HNC patients at any stage of diagnosis (Stages 0-IV);
   * Over 18 years old;
   * English and/or Spanish speaking;
   * Medically underserved, as defined by at least one or several of the following:

     1. Low-income: Below 400% of the 2016 Federal poverty levels;
     2. Uninsured: No health insurance (public or private insurance);
     3. Underinsured: e.g.: Public insurance (Medicaid, Medicare exclusive, VA); and/or 10% of annual income on out-of-pocket medical expenses for individuals below 200% of the 2016 Federal poverty levels.

   Exclusion Criteria:
   * Individuals who do not meet eligibility criteria, including individuals who do not speak English or Spanish;
   * Those who refuse treatment at one of three hospital sites;
   * Decisionally-challenged adults with cognitive or personality impairment;
   * Suicidal ideation, or
   * Intoxication (alcohol or drugs) that might interfere with their ability to consent or participate in the study;
   * Individuals from vulnerable populations (e.g., inmates or individuals on probation,
   * homeless,
   * pregnant women, and
   * those with auditory impairment.

   Note: Individuals who become pregnant or develop auditory impairments after they have been randomized to study condition may remain in the study until completion.
2. Caregivers of LC and/or HNC patients

Inclusion Criteria:

* Primary caregiver of a newly diagnosed LC and/or HNC patient (per criteria for patients);
* Over 18 years old;
* English and/or Spanish speaking;
* Medically underserved, as defined by at least one or several of the following:

  1. Low-income: Below 400% of the 2016 Federal poverty levels;
  2. Uninsured: No health insurance (public or private insurance);
  3. Underinsured:
* (c.1) Public insurance (i.e., Medicaid, Medicare exclusive, VA);
* (c.2) 10% of annual income spent on out-of-pocket medical expenses for individuals below 200% of the 2016 Federal poverty level.

Exclusion criteria:

* Individuals who do not meet eligibility criteria, including individuals who do not speak English or Spanish [at the discretion of the Site Coordinators upon recruitment];
* Caregivers of patients who refuse treatment at one of three hospital sites.
* Decisionally challenged adults with:

  1. cognitive or personality impairment,
  2. suicidal ideation, or
  3. intoxication (alcohol or drugs) that might interfere with their ability to consent or participate in the study [at the discretion of the Site Coordinators upon recruitment or the Counselor during the intervention];
* Individuals from:

  1. vulnerable populations (e.g., inmates or individuals on probation, homeless,
  2. pregnant women, and
  3. those with auditory impairment [at the discretion of the Site Coordinators upon recruitment]).
  4. Individuals who become pregnant or develop auditory impairments after they have been randomized to study condition may remain in the study until completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelinn A Borrayo, PhD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - Denver Health Medical Center, Denver, Colorado
  - University of Colorado Denver, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - Saint Joseph Hospital, Denver, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borrayo EA, Juarez-Colunga E, Kilbourn K, Waxmonsky J, Jacobson M, Okuyama S, Swaney R, Wamboldt FS, Karam S, Lopez Alvarez S, Jin X, Nguyen J. Stepped-care to improve mental health outcomes among underserved patients with lung and head and neck cancer. Psychooncology. 2023 Nov;32(11):1718-1726. doi: 10.1002/pon.6223. Epub 2023 Sep 29. PMID 37772984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Both patients and caregivers were recruited for this study. Primary outcomes data were focused on patients. Caregiver data were included as secondary analyses.
Groups:
- Patients in Enhanced Usual Care: Patients who were randomized to Enhanced Usual Care
- Patients in Stepped Care Intervention: Patients who were randomized to the Stepped Care Intervention
- Caregivers in Enhanced Usual Care: Caregivers who were randomized into Enhanced Usual Care
- Caregivers in Stepped Care Intervention: Caregivers who were randomized to the Stepped Care Intervention
Period: Baseline
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Started | 139 | 147 | 118 | 131
Completed | 123 | 120 | 107 | 97
Not Completed | 16 | 27 | 11 | 34
Not completed — Death | 5 | 8 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 4 | 10
Not completed — Lost to Follow-up | 9 | 11 | 6 | 24
Period: 6-week Follow-up
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Started | 123 (Anyone who had at least 1 follow-up after baseline.) | 120 | 107 | 97
Completed | 120 | 107 | 103 | 88
Not Completed | 3 | 13 | 4 | 9
Not completed — Death | 1 | 4 | 0 | 0
Not completed — Lost to Follow-up | 2 | 7 | 4 | 8
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Period: 3-month Follow-up and 6-month Follow-up
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Started | 120 | 107 | 103 | 88
Completed | 108 | 96 | 95 | 81
Not Completed | 12 | 11 | 8 | 7
Not completed — Death | 6 | 4 | 0 | 0
Not completed — Lost to Follow-up | 6 | 7 | 8 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Caregivers in Enhanced Usual Care: Caregivers who were randomized to Enhanced Usual Care
- Total: Total of all reporting groups
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention | Total
Number analyzed (Participants) | 139 | 147 | 118 | 131 | 535
Age, Customized [Count of Participants; unit: Participants]
  Under 18 | 0 | 0 | 0 | 0 | 0
  18 to 65 | 65 | 69 | 64 | 69 | 267
  Above 65 | 74 | 78 | 33 | 36 | 221
  Unknown or Not Report | 0 | 0 | 21 | 26 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 65 | 92 | 99 | 310
  Male | 85 | 82 | 26 | 32 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 34 | 28 | 37 | 126
  Not Hispanic or Latino | 112 | 113 | 89 | 94 | 408
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 1 | 3 | 8
  Asian | 1 | 1 | 6 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 3 | 0 | 4
  Black or African American | 6 | 9 | 3 | 7 | 25
  White | 123 | 122 | 99 | 107 | 451
  More than one race | 2 | 1 | 2 | 2 | 7
  Unknown or Not Reported | 5 | 11 | 4 | 7 | 27
Region of Enrollment [Number; unit: participants]
  United States | 139 | 147 | 118 | 131 | 286
Language Preference [Count of Participants; unit: Participants]
  English | 133 | 132 | 111 | 118 | 494
  Spanish | 6 | 15 | 7 | 13 | 41
Diagnosis [Count of Participants; unit: Participants] — Population: Diagnosis data were not collected from caregivers.
  Participants
    number analyzed (Participants) | 139 | 147 | 0 | 0 | 286
    Head and neck cancer | 60 | 60 | 0 | 0 | 120
    Lung cancer | 79 | 87 | 0 | 0 | 166
Cancer Stage [Count of Participants; unit: Participants] — Cancer Stage were clinically diagnosed by medical oncologists at each site and were self-reported by patients in the baseline survey. The cancer stages varied between stage 0, I, II, III, and IV with IV being the most advanced. Population: No cancer stage was collected from the caregivers.
  Participants
    number analyzed (Participants) | 139 | 147 | 0 | 0 | 286
    Stage 0, I, & II | 65 | 67 | 0 | 0 | 132
    Stage III & IV | 73 | 78 | 0 | 0 | 151
    Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Step at Baseline [Count of Participants; unit: Participants] — The treatment steps that participants were assigned to, based on their personal level of distress included:
  Step 1: Watchful Waiting Step 2: Self-Help Guide Step 3: Coping Skills Training Step 4: Cognitive-Behavioral Therapy
  Participants
    Step 1 & 2 | 106 | 114 | 89 | 106 | 415
    Step 3 & 4 | 33 | 32 | 29 | 25 | 119
    Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Symptoms of Depression-Patients
Description: Patient-Reported Outcomes Measurement Information System (PROMIS)-Cancer (CA) Form v1.0 - Depression (30 items). The range is from 8 to 40. Higher score indicates worse outcome (higher depression). Raw scores were used in analyses.
Time Frame: 6-months
Population: Intention to treat population- all participants who were randomized were included in this analysis. The reported means correspond to the observed means at 6 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention
Number analyzed (Participants) | 139 | 147
score on a scale | 15.3 (7.0) | 13.2 (5.7)
Statistical Analysis 1: Comparison: Patients in Enhanced Usual Care vs Patients in Stepped Care Intervention; A linear mixed model (LMM) with random intercepts for both patients and clinics has been used, with adjustment for cancer type and cancer stage. The study was powered for testing the hypothesis of no group differences in change over the four time points (baseline, 6-weeks, 3-months and 6-months). A significant group by time interaction was hypothesized; Test type: Superiority; p = 0.0057, Mixed Models Analysis — Since there are three primary outcomes (depression, anxiety and coping scores) in the study, the significance level was set a priori at 0.0167 (alpha = 0.05/3); The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 1.75, 95% CI 2-sided [0.52 to 2.98] — The estimate represents the difference in expected means at the 6-month time point between the intervention and usual care arms

2. Primary Outcome: Symptoms of Anxiety-Patients
Description: Patient-Reported Outcomes Measurement Information System, Anxiety (PROMIS-Ca) Form v1.0- Anxiety (22 items). The range of scores is between 8 and 40. The raw scores were used. Higher score corresponds to worse outcome.
Time Frame: 6-months
Population: Intention to treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Stepped-Care Intervention
Number analyzed (Participants) | 139 | 147
score on a scale | 16.0 (7.0) | 13.9 (6.6)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Stepped-Care Intervention; Linear mixed models (LMM) have been used with time and the interaction between time and group as fixed effects. A structure of random effects that includes random intercepts for patients was used. The study was powered for testing the hypothesis of no group differences in change over the four time points. A significant group by time interaction was hypothesized; Test type: Superiority; p = 0.0243, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 1.46, 95% CI 2-sided [0.19 to 2.73] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in Coping-Patients
Description: Coping Self-Efficacy (26 items). Scores can rage from 0 to 260. Higher score corresponds to better outcome.
Time Frame: 6-months
Population: Intention to treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Stepped-Care Intervention
Number analyzed (Participants) | 139 | 147
score on a scale | 190 (55) | 207 (54)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Stepped-Care Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0061, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of an interaction between time and intervention arm; Mean Difference (Final Values) = -15.31, 95% CI 2-sided [-26.23 to -4.39] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Coping-Caregivers
Description: Coping Self-Efficacy (26 items). Higher score corresponds to better outcome. Scores can rage from 0 to 260.
  The number of caregivers randomized and analyzed was 118 and 131 in the enhanced usual care and intervention groups, respectively.
Time Frame: 6-months
Population: Intention to treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Usual Care | Stepped-Care Intervention
Number analyzed (Participants) | 118 | 131
score on a scale | 192 (52) | 211 (50)
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Stepped-Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.21, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = -7.73, 95% CI 2-sided [-19.73 to 4.27] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Symptoms of Anxiety-Caregivers
Description: PROMIS Form v1.0 - Anxiety (29 items). The range of scores is from 8 to 40. Higher score indicates worse outcome (higher anxiety). Raw scores were used in analyses.
  The number of caregivers randomized and analyzed was 118 and 131 in the enhanced usual care and intervention groups, respectively.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Number analyzed (Participants) | 118 | 131
score on a scale | 17 (7) | 14 (7)
Statistical Analysis 1: Comparison: Caregivers in Enhanced Usual Care vs Caregivers in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.052, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 1.52, 95% CI 2-sided [-0.01 to 3.05] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Symptoms of Depression-Caregivers
Description: PROMIS Form v1.0 - Depression (28 items). The range is from 8 to 40. Higher score indicates worse outcome (higher depression). Raw scores were used in analyses.
  The number of caregivers randomized and analyzed was 118 and 131 in the enhanced usual care and intervention groups, respectively.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Number analyzed (Participants) | 118 | 131
score on a scale | 15.0 (6.9) | 13.2 (5.7)
Statistical Analysis 1: Comparison: Caregivers in Enhanced Usual Care vs Caregivers in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.214, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 0.91, 95% CI 2-sided [-0.52 to 2.36] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Health-Related Quality of Life-Patients
Description: FACT-G version 4 (27 items). The range is 0-108. Higher values indicate better QOL.
Time Frame: 6-months
Population: Intention to treat population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention
Number analyzed (Participants) | 139 | 147
score on a scale | 73 (19) | 80 (19)
Statistical Analysis 1: Comparison: Patients in Enhanced Usual Care vs Patients in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0134, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = -4.16, 95% CI 2-sided [-7.45 to -0.87] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Perceived Stress-Patients
Description: Perceived Stress Scale (PSS) (14 items). The range of scores is 0-40. Higher values indicate higher stress.
Time Frame: 6-months
Population: intention to treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention
Number analyzed (Participants) | 139 | 147
score on a scale | 14 (7) | 13 (7)
Statistical Analysis 1: Comparison: Patients in Enhanced Usual Care vs Patients in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.42, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-0.9 to 2.12] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Perceived Stress-Caregivers
Description: Perceived Stress Scale (PSS) (14 items). The range is from 0 to 40. Higher values indicate higher stress.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Number analyzed (Participants) | 118 | 131
score on a scale | 15 (7) | 11 (7)
Statistical Analysis 1: Comparison: Caregivers in Enhanced Usual Care vs Caregivers in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0269, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 1.77, 95% CI 2-sided [0.2 to 3.34] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Caregiving Burden-Caregivers
Description: Zarit Burden Interview (ZBI) (12 items). The range of scores is 0-48. Higher scores represent higher burden.
Time Frame: 6-months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
Number analyzed (Participants) | 118 | 131
score on a scale | 13 (9) | 9 (8)
Statistical Analysis 1: Comparison: Caregivers in Enhanced Usual Care vs Caregivers in Stepped Care Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0044, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; The pvalue corresponds to the hypothesis of the interaction effect between time and group (intervention arm); Mean Difference (Final Values) = 2.56, 95% CI 2-sided [0.8 to 4.32] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Between baseline through the six month follow-up. Adverse events can be reported by the study coordinators at anytime from baseline through completion of the 6 month follow-up.
Arm/Group | Patients in Enhanced Usual Care | Patients in Stepped Care Intervention | Caregivers in Enhanced Usual Care | Caregivers in Stepped Care Intervention
All-Cause Mortality (participants affected / at risk) | 13/139 | 18/147 | 1/118 | 0/131
Serious Adverse Events (participants affected / at risk) | 13/139 | 19/147 | 1/118 | 0/131
Other Adverse Events (participants affected / at risk) | 0/139 | 0/147 | 0/118 | 0/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients in Enhanced Usual Care (N=139) | Patients in Stepped Care Intervention (N=147) | Caregivers in Enhanced Usual Care (N=118) | Caregivers in Stepped Care Intervention (N=131)
Death (General disorders) | 13 (13) | 18 (18) | 1 (1) | 0 (0) — Head-and-neck/lung cancer or complications related to the diagnoses
Respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03016403/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT03016403/ICF_001.pdf